CLINICAL TRIAL: NCT04725383
Title: Amitriptyline for Repetitive Behaviors in Children and Adolescents With Autism Spectrum Disorders
Brief Title: Amitriptyline for Repetitive Behaviors in Autism Spectrum Disorders
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The PI is retiring.
Sponsor: University of Missouri, Kansas City (Other)
Responsible Party: Principal Investigator, Jessica Hellings, Professor of Psychiatry, University of Missouri, Kansas City
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015984; 17-055 (Other: Truman Medical Center)
Record Dates: First submitted 2021-01-07; First posted 2021-01-26 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorder; Repetitive Compulsive Behavior
Keywords: amitriptyline; autism; repetitive behaviors
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Amitriptyline

STUDY DESIGN:
Intervention Model Description: Randomized double-blind placebo-controlled clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All individuals involved in the study will be blinded as to drug or placebo condition, except for one psychiatry co-investigator who will remain unblinded and check that amitriptyline levels are not above the maximum for the laboratory therapeutic range.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- amitriptyline (Active Comparator): Subjects will receive active amitriptyline compounded into look-alike capsules to resemble placebo capsules. Dosing will be as tolerated, up to tid and maximum of 100mg/day or 1.5mg/kg/day, for 10 weeks.
  Interventions: Drug: amitriptyline
- placebo (Placebo Comparator): Subjects in this arm will receive placebo compounded into capsules that resemble the compounded amitriptyline capsules, up to 4 capsules a day (1 qam, 1 q4pm and 2 capsules qhs), for 10 weeks.
  Interventions: Drug: amitriptyline

INTERVENTIONS:
Drug: amitriptyline — Amitriptyline is a tricyclic antidepressant being studied off-label here for repetitive behaviors in autism spectrum disorders.
  Other Names: Elavil

SUMMARY:
The investigators will recruit 30 children and adolescents (15 per group x 2 groups) aged 6 to 17 years with ASD and significant repetitive behaviors that cause problems to them and to others around them. Subjects will be randomized to either amitriptyline (AMI), dosed flexibly according to response and tolerability with a maximum dose of 100mg per day or 1.5mg/kg/day, in divided doses to minimize side effects, or placebo in look-alike capsules, for 10 weeks. Rating scales will be used to measure outcomes.

DETAILED DESCRIPTION:
At the screening visit, investigators will perform a full history-taking, mental status examination, physical and neurological examinations, the ADI-R with a caregiver or parent to confirm autism, an EKG and complete rating scales, as well as a pregnancy test (beta-HCG) in sexually active females of childbearing age. Sexually active females of childbearing age must be on a form of birth control during the study, such as the oral contraceptive pill, intrauterine device or Depo Provera shot. A parent or guardian will sign informed consent, as appropriate, and written assent will be obtained from subjects. Blood tests for CBC and diff, CMP, amitriptyline level will be obtained at at baseline (except for amitriptyline) week 6 and 10.

Subjects will be randomized to amitriptyline (AMI) or placebo. Parents and guardians will be instructed to lock up all medications, warned regarding overdose toxicity and this will be documented in writing. Treatment will be low dose AMI or placebo for 12 weeks. Study visits will occur at weeks 0,1, 2, 3, 4, 5, 6, 8, and 10.

Investigators will complete a Clinical Global Impressions scale (CGI), and have the accompanying adult or parent complete rating scales, at each visit, notably the Child Yale Brown Obsessive Compulsive scale modified for Pervasive Developmental Disorder (CYBOCS-PDD), Aberrant Behavior Checklist-Irritability subscale (ABC-I), Repetitive Behavior Scale-Revised (RBS-R), ADHD-RS, adverse events form, ADI-R item 11 for phrase speech, and a concomitant treatment review form, which will also detail for example any over-the-counter medications, supplements or antibiotics taken. Also a gastrointestinal symptom form based on that used by Valicenti-McDermott et al. 2008.

At all interim visits, the PI will perform a follow-up history taking, mental status examination, vital signs, rating scales as above and study drug dispensing. Any unused capsules must be returned at each visit, to monitor compliance as well as to prevent accidental overdose. Parents and caregivers will agree to lock medication up, and will be reminded of overdose toxicity at each study visit, with written documentation.

Flexible dosing, arranged by calling the pharmacy to randomize the subject and then dispense and mail study capsules, according to the psychiatrist's instructions at each visit, to a maximum dose of 100mg/day or 1.5mg/kg/day maximum by subject weight.

Individuals and their parents or guardians will be questioned about suicidal ideation at each visit, and instructed to call study staff if that should arise. At that time the PI will arrange an urgent visit to closely assess risks of remaining in the study. In our experience suicidal ideation has not occurred. Subjects may drop out at any time however, and in the unlikely case, if warranted, be admitted to hospital for close observation.

The study will be double- blind and placebo-controlled. All investigators except a psychiatry co-investigator will be blinded, as will caregivers, families and subjects.

ELIGIBILITY:
Inclusion Criteria:

* males and females
* ages 6-17 years;
* diagnosis of ASD validated by the Autism Diagnostic Interview- Revised (Lord et al. 1994); CGI-S rating of at least Moderate problem CYBOCS-PDD score of at least 8 or more for compulsive behaviors (sum of items 1A, 2, 3 and 5)
* Intellectual Disability if present to be no greater than moderate by history (ie IQ>35).

Exclusion Criteria:

* unable to complete an EKG recording, even with low dose risperidone and alprazolam if needed an hour before, and repeated at the time (if needed), of the procedure,
* QTc on EKG of 440 or more
* absence of a reliable caregiver
* amitriptyline allergy
* previous neuroleptic malignant syndrome
* seizures in the past 3 months
* bipolar mood disorder
* current or past psychosis
* unstable medical illness
* previous adequate trial of amitriptyline
* using other psychotropic medications apart from melatonin for sleep or lorazepam 1mg as needed up to once a day for severe outbursts.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impressions scale-Improvement of Much Improved (2) or Very Much Improved (1) | up to 10 weeks
  1 Very Much Improved to 7 Very Much Worse
Child Yale Brown Obsessive Compulsive Scale- Pervasive Developmental Disorders (CYBOCS-PDD) | up to 10 weeks
  0-20; high scores are more severe

SECONDARY OUTCOMES:
Repetitive Behavior Scale-revised | up to week 10
  0-129; high scores are more severe

OTHER OUTCOMES:
Social Responsiveness scale-2 | Baseline, week 10
  34-90; high scores are more severe
Attention-Deficit-Hyperactivity Disorder Rating Scale-Revised IV | up to week 10
  0-54; high scores are more severe
Aberrant Behavior Checklist-Irritability subscale | up to week 10
  0-45; high scores are more severe
ADI-R Item 16 for social vocalization/chat | baseline, week 6 and 10
  0-3; highest scores indicate poorest

CONTACTS AND LOCATIONS:
Overall Officials: Jessica A. Hellings, MD, Principal Investigator — University of Kansas City-Missouri and Truman Behavioral Health
Locations (1):
- University Health Behavioral Health Canvas Building, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhatti I, Thome A, Smith PO, Cook-Wiens G, Yeh HW, Gaffney GR, Hellings JA. A retrospective study of amitriptyline in youth with autism spectrum disorders. J Autism Dev Disord. 2013 May;43(5):1017-27. doi: 10.1007/s10803-012-1647-0. PMID 23135317